CLINICAL TRIAL: NCT05889156
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled 28- Day Phase II Proof of Concept Study to Evaluate the Efficacy and Safety of NST-1024 400 mg BID Versus Placebo in Statin-Naïve or Statin-Stable Hypertriglyceridemic Subjects
Brief Title: Study of the Efficacy and Safety of NST-1024 Versus Placebo in Subjects With Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NST-1024-03
Record Dates: First submitted 2023-03-16; First posted 2023-06-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: High Triglycerides
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matched Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- NST-1024 (Active Comparator): NST-1024 400 mg BID
  Interventions: Drug: NST-1024

INTERVENTIONS:
Drug: NST-1024 — 400 mg BID
  Arms: NST-1024
Other: Placebo — matched placebo to active arm
  Arms: Matched Placebo

SUMMARY:
This is a Phase IIa,multicentre proof of concept study consisting of 2 study periods to study Treatment with NST-1024 as an adjunct to diet to reduce triglyceride (TG) levels in subjects with TG levels of ≥500 mg/dL and ≤2000 mg/dL; determined by percentage change in TG from baseline after 28 days of treatment.

The two periods consist of:

1. A 3-week screening period that includes a TG qualifying period, and
2. A 28-days, double-blind, randomized, parallel group, placebo-controlled treatment period.

Subjects will return to the study site for a follow-up visit 2 weeks after the last dose.

Approximately 50 subjects will be randomized at approximately 15-35 centers in USA.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding of the study procedures, willing to adhere to the study schedules, and agreement to participate in the study by giving written informed consent prior to screening (Visit 1 Week -3]) assessments;
2. Men or women 18 to 79 years of age, inclusive;
3. If on statin or non-statin lipid-altering therapy, such as ezetimibe, niacin >200 mg/day, bempedoic acid, fibrates, prescription omega-3 products, other consumer products containing omega-3 fatty acids, or other herbal products or dietary supplements with potential lipid and glucose-altering effects, subject's use must be stable for ≥28 days prior to the first TG baseline qualifying measurement (i.e., Visit 1 [Week -3]), and should remain stable thereafter for the duration of study participation;
4. Fasting TG levels ≥500 mg/dL and ≤2000 mg/dL (based on an average [arithmetic mean] of Visit 1 and Visit 2). Note: In cases in which a subject's average TG level from Visit 1 and Visit 2 falls outside the range for entry into the study, an additional visit (Visit 2a) can be arranged up to 7 days after Visit 2 for an additional measurement of fasting TG levels. If a third sample is collected, entry into the double-blind treatment period will be based on the average of the highest TG value from Visit 1 and 2 and the Visit 2a value. Neither one of the two values used for the arithmetic mean can be less than 400 mg/dL;
5. If using oral or injectable weight loss drug, subjects must maintain stable dose of all oral and injectable weight loss drugs (e.g., GLP-1 receptor agonists) for at least 3 months prior to screening (i.e., Visit 1 [Week -3]), and during participation in the study.
6. Willingness to maintain stable diet and physical activity level throughout the study
7. If a smoker, no plans to change smoking habits during the study period.
8. Agree to use appropriate contraceptive methods based on biological sex and child-bearing potential as outlined in Section 12.5 of the protocol.
9. Agree to abstain from sperm or egg donation through 90 or 30 days, respectively, after administration of the last dose of IP.

Exclusion Criteria:

1. Body mass index >50 kg/m2;
2. Participation in another clinical study involving an investigational agent within 30 days prior to screening or 5½ half-lives whichever is longer (Visit 1 [Week -3]);
3. Type 1 diabetes mellitus;
4. HbA1c > 9.5% at screening (Visit 1 [Week -3]);
5. History of stroke, myocardial infarction, life-threatening arrhythmia, or coronary revascularization within 6 months prior to screening;
6. History of chronic pancreatitis or acute pancreatitis in the last year. Subjects at risk of developing pancreatitis (e.g., known cholelithiasis, known alcohol abuse or multiple incidences of acute pancreatitis) per the PI's assessment are excluded. Subjects with a history of acute pancreatitis due to gallstones who have been treated with cholecystectomy are allowed.
7. History of symptomatic gallstone disease unless treated with cholecystectomy;
8. History of nephrotic range (>3 g/day) proteinuria;
9. Estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73 m2
10. QTcF interval of >450ms for males or >470ms for females
11. A history of additional risk factors for torsades de pointes (TdP) (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)
12. The use of concomitant medications that prolong the QT/QTc interval (Table 1);
13. History or evidence of major and clinically significant hepatic, pulmonary, renal, hematologic, gastrointestinal (including clinically significant malabsorption), endocrine, immunologic, dermatologic, neurologic, psychiatric, oncologic, or allergic (including drug allergies, but excluding untreated or treated seasonal allergies at the time of dosing) disease that would interfere with the conduct of the study or interpretation of the data;
14. Known lipoprotein lipase impairment or deficiency (Fredrickson Type I), apolipoprotein C-II deficiency, or familial dysbetalipoproteinemia (Fredrickson Type III);
15. Requirement for peritoneal dialysis or haemodialysis for renal insufficiency;
16. History of malignancy, unless:

    I. All treatment for the malignancy was completed ≥2 years prior to screening and there is no evidence of disease; II. Curatively resected squamous or basal cell carcinomas of the skin, carcinomas in situ of the cervix or uterus, ductal breast cancer in situ or low-grade prostate cancer III. Squamous cell or basal cell skin carcinomas that are not requiring tumour directed treatment during the subject's participation in the study
17. History of bariatric surgery less than 2 years prior to randomization. A history of bariatric surgery utilizing the gastric bypass technique (Roux-en-Y) or biliopancreatic diversion with duodenal switch is exclusionary;
18. Uncontrolled hypertension;
19. Known to be infected with human immunodeficiency virus (HIV) AND who are not on stable antiretroviral therapy OR have a confirmed plasma HIV-1 RNA (Viral Load) > lower limit of detection despite antiretroviral therapy OR have a CD4+ T-cell count <350 cell/μL OR a history of acquired immunodeficiency syndrome(AIDS);
20. Hepatitis B or C:

    I. Acute or chronic Hepatitis B infection based on a positive hepatitis B surface antigen (HBsAg) test at screening (Visit 1 [Week -3]). Subjects with a past hepatitis B virus (HBV) infection or resolved HBV infection (defined by presence of hepatitis B core antibody (HBcAb) and absence of HbsAg are eligible if confirmed with negative HBV DNA test performed at screening; II. Positive test for hepatitis C antibody at screening (Visit 1 [Week -3]), except for those who have been successfully treated for hepatitis C infection and have achieved sustained virologic response for ≥1 year and who have a negative reflex HCV RNA test;
21. Anticipation of major surgery during the screening or double-blind treatment periods of the study;
22. Treatment with chronic prescription pharmacotherapy for metabolic or CV disease management or risk factor modification (e.g., antihypertensive and antidiabetic medications) that has not been stable for ≥28 days prior to screening (Visit 1 [Week -3]);
23. Ongoing treatment with cyclophosphamide (unless chronic oral administration for inflammatory conditions such as rheumatoid arthritis or inflammatory bowel disease), or isotretinoin;
24. Treatment with tamoxifen, estrogens, or progestins that has not been stable for ≥28 days prior to screening (Visit 1 [Week -3]);
25. Use of systemic corticosteroids at a dose >7.5mg daily prednisolone equivalent (per Appendix A) ≤28 days prior to screening or anticipated use during study. Use of local injectable, inhaled, nasal administration, topical corticosteroids, or low dose glucocorticoids (≤7.5 mg prednisolone equivalent) is permitted. Low dose oral glucocorticoids should have been used for ≥ 3 months and stable for ≥ 28 days prior to baseline (Visit 3);
26. Thyroid-stimulating hormone (TSH) > 2.0 x upper limit of normal (ULN), clinical evidence of hypothyroidism, or thyroid hormone therapy that has not been stable for ≥6 weeks prior to screening (Visit 1 [Week -3]);
27. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x ULN, unless exercise-related;
28. Unexplained CK concentration >5 × ULN or CK elevation due to known muscle disease (e.g., polymyositis, mitochondrial dysfunction);
29. Other recent or current serious disease that may interfere with the conduct of the study (renal, ophthalmic, pulmonary, hepatic, biliary, gastrointestinal, mental disorder, infectious disease, or cancer);
30. Blood donation of ≥1 pint (0.5 L) within 8 weeks prior to screening (Visit 1 [Week -3]) or anticipated blood donation during study, or plasma donation within 7 days prior to screening (Visit 1 [Week -3]);
31. History of illicit drug use or alcohol abuse within 1 year of screening (Visit 1 [Week -3]). Alcohol abuse is defined as >21 standard drinks per week in men and >14 standard drinks per week in women, on average;
32. Any condition or therapy, which, in the opinion of the investigator, might pose a risk to the subject or make participation in the study not in the subject's best interest;
33. Poor mental function or any other reason to expect subject difficulty in complying with the requirements of the study; or in the investigator's opinion, not able to comply with study procedures.
34. Pregnancy or breastfeeding.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of NST-1024 by percentage change in TG | 4 weeks
  Evaluate the efficacy of NST-1024 400 mg BID by assessment of the percentage change in TG from baseline after 28 days of treatment

SECONDARY OUTCOMES:
Percent Change in Cholesterol Values | 4 weeks
  Percent changes in TC, HDL-C, LDL-C, calculated. non-HDL-C, and VLDL-C from baseline to Week 4
Percent change in Apolipoprotein B and Apolipoprotein C3 | 4 weeks
  Percent changes in ApoB and ApoC3 from baseline to Week 4.
Percent Change in Lipoprotein a | 4 weeks
  Percent change in Lp(a) from baseline to Week 4.
Percent Change in remnant-like particle cholesterol (RLP-C) | 4 weeks
  Percent Change in RLP-C from baseline to Week 4.
Changes in fasting plasma glucose, fasting plasma insulin, and HbA1c | 4 weeks
  Changes in fasting plasma glucose (FPG), fasting plasma insulin (FPI) and HbA1c from baseline to Week 4
Change in insulin resistance. | 4 weeks
  Change in insulin resistance, as assessed by the homeostasis model index insulin resistance, from baseline to Week 4
Change in lipoprotein associated phospholipase A2 | 4 weeks
  Percent change in lipoprotein associated phospholipase A2 from baseline to Week 4
Change in hsCRP | 4 weeks
  Change in hsCRP from baseline to Week 4
Safety Assessments | ~ 8 weeks
  Incidence of Treatment-Emergent Adverse Events and abnormalities in clinical laboratory measurements (chemistry, haematology, and urinalysis), 12-lead ECGs, blood pressure, and physical examinations will be evaluated and monitored for any safety events through the study duration from screening through follow up.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - University of Alabama - Heersink School of Medicine, Birmingham, Alabama
  - Alliance for Multispecialty Research, LLC (AMR) - Daphne, Daphne, Alabama
  - Alliance for Multispecialty Research, LLC (AMR) - Phoenix, Tempe, Arizona
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Velocity Clinical Research - Costal Heart, Santa Ana, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Velocity Clinical Research, New Smyrna Beach, Edgewater, Florida
  - Clearwater Cardiovascular Consultants, Largo, Florida
  - Floridian Clinical Research, Miami Lakes, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Lifeline Primary Care/ CCT Research, Lilburn, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Deaconess Clinic - Indiana, Evansville, Indiana
  - Velocity Clinical Research, Valparaiso, Valparaiso, Indiana
  - Alliance for Multispecialty Research, LLC (AMR) - Newton, Newton, Kansas
  - University of Louisville - UoL Physicians Outpatient Center, Louisville, Kentucky
  - Troy Internal Medicine, Troy, Michigan
  - Clay Platte Family Medicine / CCT Research, Kansas City, Missouri
  - Velocity Clinical Research - Kearney, Lincoln, Nebraska
  - Cenexel HRI, Berlin, New Jersey
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Velocity Clinical Research - Cleveland, Cleveland, Ohio
  - Hatboro Medical Associates/ CCT Research, Hatboro, Pennsylvania
  - Mercado Medical Practice / CCT Research, Philadelphia, Pennsylvania
  - Palmetto Clinical Reserach, Summerville, South Carolina
  - Velocity Clinical Research - Union, Union, South Carolina
  - Apex Mobile Clinical Research, Bellaire, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Ogden Clinic, Mount View/CCT Research, Pleasant View, Utah
  - Velocity Clinical Research - Salt Lake City, Salt Lake City, Utah